CLINICAL TRIAL: NCT03395535
Title: Health-Related Quality of Life in Two Pathways for Newly Diagnosed Open Angle Glaucoma and Ocular Hypertension: an Unmasked, Multi-centre, Randomised Controlled Trial of Initial Selective Laser Trabeculoplasty Versus Medical Therapy
Brief Title: Laser-1st vs Drops-1st for Glaucoma and Ocular Hypertension
Acronym: LIGHT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mr Gus Gazzard, CONSULTANT OPHTHALMOLOGIST, Moorfields Eye Hospital NHS Foundation Trust
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: GAZG1001; HTA 09/104/40 - LiGHT (Other: NIHR HTA); ISRCTN 32038223 (Other: ISRCTN)
Record Dates: First submitted 2013-05-24; First posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: Primary Open Angle Glaucoma; Glaucoma; Ocular Hypertension; POAG; SLT; Laser
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All clinical tests and outcomes are by masked observers.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 'Laser-1st' (Experimental): Initial Selective Laser Trabeculoplasty (SLT) [PROCEDURE] followed by conventional medical therapy (eye-drops) as required.
  All participants in this arm start their treatment pathway with SLT. If this does not reach the predefined, patient-specific target IOP then repeat laser (once only) is given. If the IOP target is then not reached additional treatment with all standard medications may be used and ultimately surgery (trabeculectomy with mitomycin C) as needed.
  Interventions: Procedure: Primary Selective Laser Trabeculoplasty Treatment Pathway
- Medicine-1st (Active Comparator): Conventional medical therapy [DRUG] without laser. All participants in this arm start their treatment pathway medical treatment. If the IOP target is then not reached, additional treatment with all standard medications may be used and ultimately surgery (trabeculectomy with mitomycin C) as needed.
  During this pathway of treatment all commercially available medical treatments (eye-drops) are permitted according to a pre-specified step-wise intervention protocol described in detail in the publicly available trial protocol. This begins with prostaglandin analogues, then beta-blockers followed by alpha agonists or carbonic anhydrase inhibitors. The full range of available doses, treatments and drugs is beyond this short summary.
  Interventions: Drug: Primary Medical Treatment Pathway

INTERVENTIONS:
Procedure: Primary Selective Laser Trabeculoplasty Treatment Pathway — Primary Selective Laser Trabeculoplasty Treatment (followed by medications as required) Pathway.
  First treatment is SLT, 100 shots of laser over 360 degrees. If this does not reach the target IOP then repeat laser (once only) is given. If IOP not at target additional treatment with all standard medications may be used and ultimately surgery (trabeculectomy ).
  All available medical treatments (eye-drops) are permitted according to a pre-specified intervention protocol described in detail in the publicly available trial protocol. This begins with prostaglandin analogues, then beta-blockers followed by alpha agonists or carbonic anhydrase inhibitors. The full range of available doses, treatments and drugs is beyond this short summary.
  Other Names: SLT; "Laser First"
  Arms: 'Laser-1st'
Drug: Primary Medical Treatment Pathway — Primary Medical Treatment Pathway (multiple medications, as required). If IOP not at target additional treatment with all standard medications may be used and ultimately surgery (trabeculectomy ).
  All available medical treatments (eye-drops) are permitted according to a pre-specified intervention protocol described in detail in the publicly available trial protocol. This begins with prostaglandin analogues, then beta-blockers followed by alpha agonists or carbonic anhydrase inhibitors. The full range of available doses, treatments and drugs is beyond this short summary.
  Other Names: Conventional medical therapy; "Medicine First"
  Arms: Medicine-1st

SUMMARY:
This is a randomized study with two treatment arms: 'initial Selective Laser Trabeculoplasty (SLT) followed by conventional medical therapy as required' ('Laser-1st') and 'medical therapy without laser ('Medicine-1st'). It compares quality of life in the two arms at three years, while also examining the incremental cost and cost-effectiveness of Laser-1st versus Medicine-1st.

DETAILED DESCRIPTION:
Subjects are randomly allocated to one of two treatment arms that examine treatment pathways, rather than comparing single treatments alone: 'initial Selective Laser Trabeculoplasty (SLT) followed by conventional medical therapy as required' ('Laser-1st') and 'medical therapy without laser ('Medicine-1st'). We compare quality of life in the two pathways (arms) over three years, while also examining the incremental cost and cost-effectiveness of Laser-1st versus Medicine-1st.

A 'Treat in Pursuit of Control' design (TPC) compares two different routes to a pre-defined target Intraocular pressure (IOP) (pathways). It is a pragmatic study that uses published guidelines to make the complex clinical treatment choices faced in managing glaucoma, standardised between treatment arms by use of computer treatment algorithms. A UK National Institute for Health and care Excellence (NICE)-compliant evidence-based IOP Treatment Target 1 is set for each patient, according to the study treatment algorithms. They then proceed through stepped increments of treatment intensity (up to and including surgery) until a predetermined Target IOP is reached. Target IOP is reassessed in the light of objective clinical evidence of stability of glaucomatous optic neuropathy (GON) and visual function using visual field tests and automated optic nerve evaluation. Health Related Quality of Life (HRQL) and secondary outcomes are compared for patients in each pathway.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open angle glaucoma (defined as an open drainage angle and reproducible glaucomatous visual field defects as tested by the Swedish Interactive Threshold Algorithm (SITA) algorithm on the Humphrey Visual Field or glaucomatous optic neuropathy)
* OR
* Ocular hypertension (intra-ocular pressure above 21mmHg and requiring treatment as per National Institute of Health and Care Excellence (NICE) Guidelines).
* Able to provide informed consent.

Exclusion Criteria:

* Advanced glaucoma in the potentially eligible eye as determined by Early Manifest Treatment Guidelines (EMGT) criteria 77: visual field loss mean deviation worse than -12dB in the better or -15dB in the worse eye.
* Secondary glaucoma (e.g. pigment dispersion syndrome, rubeosis, trauma etc) or any angle closure.
* Any contra-indication to selective laser trabeculoplasty (e.g. unable to sit at the laser-mounted slit-lamp; past history of uveitis).
* Unable to use topical medical therapy due to e.g. physical infirmity and a lack of carers able to administer daily eye-drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 718 (Actual)
Dates: Start 2012-10-01; Primary Completion 2017-12-25 (Actual); Study Completion 2017-12-25 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life using EQ-5D | 3 years
  Quality Adjusted Life Years by EQ-5D health states

SECONDARY OUTCOMES:
Health Related Quality of Life using GUI | 3 years
  Glaucoma-specific treatment-related quality of life: Glaucoma Utility Index (GUI)
Cost-effectiveness ratio | 3 years
  Incremental Cost Effectiveness Ratio
Cost-effectiveness | 3 years
  Cost per Quality Adjusted Life Year (QALY)
Glaucoma Symptom Score (GSS) | 3 years
  Disease and treatment-related symptom score (patient reported outcome, PROM)
Glaucoma Quality of Life-15 (GQL-15) | 3 years
  Patient Reported Visual Function Score (patient reported outcome, PROM)
Glaucoma Utility Index (GUI) | 3 years
  Disease-Specific Utility Score (patient reported outcome, PROM)
Visual Acuity | 3 years
  Visual Function measured using LogMAR acuity.
Humphrey Visual Field Assessments | 3 years
  Visual Function measured using Mean Deviation
Heidelberg Retinal Tomographie optic nerve analysis | 3 years
  Optic nerve structure, measured in mean near-retinal rim width.
Goldmann Applanation Tonometry measured intra-ocular pressure | 3 years
  Clinical outcome of intra-ocular pressure lowering, mmHg.
Hospital visit frequency | 3 years
  Objective measures of treatment pathway efficacy, measured by number of hospital visits in two treatment arms over trial period.
Treatment intensity | 3 years
  Objective measures of treatment pathway efficacy, measured by number of medications used in two treatment arms over trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Gus Gazzard, MA FRCOphth, Principal Investigator — Moorfields Eye Hospital / UCL BRC
Locations (1):
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
To supply, upon request and mutually agreed terms, IPD level anonymised data where permitted by local regulations and national law.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For as long as is permissible under local regulations and national law.
Access Criteria: To Be Confirmed

REFERENCES:
- [Background] Vickerstaff V, Ambler G, Bunce C, Xing W, Gazzard G; LiGHT Trial Study Group. Statistical analysis plan for the Laser-1st versus Drops-1st for Glaucoma and Ocular Hypertension Trial (LiGHT): a multi-centre randomised controlled trial. Trials. 2015 Nov 11;16:517. doi: 10.1186/s13063-015-1047-9. PMID 26559142
- [Background] Gazzard G, Konstantakopoulou E, Garway-Heath D, Barton K, Wormald R, Morris S, Hunter R, Rubin G, Buszewicz M, Ambler G, Bunce C; LiGHT Trial Study Group. Laser in Glaucoma and Ocular Hypertension (LiGHT) trial. A multicentre, randomised controlled trial: design and methodology. Br J Ophthalmol. 2018 May;102(5):593-598. doi: 10.1136/bjophthalmol-2017-310877. Epub 2017 Sep 13. PMID 28903966
- [Background] Konstantakopoulou E, Gazzard G, Vickerstaff V, Jiang Y, Nathwani N, Hunter R, Ambler G, Bunce C; LiGHT Trial Study Group. The Laser in Glaucoma and Ocular Hypertension (LiGHT) trial. A multicentre randomised controlled trial: baseline patient characteristics. Br J Ophthalmol. 2018 May;102(5):599-603. doi: 10.1136/bjophthalmol-2017-310870. Epub 2017 Oct 5. PMID 28982956